CLINICAL TRIAL: NCT00344435
Title: Factor VIII Inhibitor Formation: Identifying Predisposing Genetic Factors
Brief Title: Genetic Susceptibility to Factor VIII Inhibitors
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905160; 05-C-N160
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-04-05

CONDITIONS: Hemophilia
Keywords: Hemophilia; Antibody; Mutations; SNP; clotting
MeSH Terms: conditions — Hemophilia A; Thrombosis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional

SUMMARY:
This international study will identify genetic factors that may influence the development of inhibitory antibodies in patients with hemophilia A after treatment with factor VIII. Bleeding episodes in patients with inhibitors are often more difficult to treat. Previous research indicates that genetic factors play a role in the development of inhibitors. A better understanding of the influence of genes in this treatment complication may be helpful in predicting, treating or preventing inhibitors.

People in families in which one or more members have severe factor VIII deficiency and one or more have a history of an inhibitor may be eligible for this study. Participants fill out a form with questions about the person's relationship to other family members taking part in the study. Those with hemophilia provide a brief medical history, including hemophilia-related information, inhibitor history and the presence of other conditions such as hepatitis C and HIV. All participants have a blood sample taken for laboratory and research tests.

DETAILED DESCRIPTION:
In collaboration with investigators of the Hemophilia Inhibitor Genetic Study (HIGS) multicenter study and the University of Lund, University Hospital, Malmo, Sweden, we propose to assess the role of genetic variants in the process of developing inhibitors to Factor VIII in persons with hemophilia. The discovery of genetic associations offers the potential to direct clinical management in order to prevent inhibitor development and improve clinical care in patients with inhibitors.

ELIGIBILITY:
* INCLUSION CRITERIA

DNA and relevant clinical data from properly consented hemophiliac subjects and family members (maximum estimated = 3500) will be provided to the LGD for genotyping and analysis.

EXCLUSION CRITERIA

No available subjects will be excluded to maximize power.

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1187 (Actual)
Dates: Start 2005-05-24; Study Completion 2016-04-05

PRIMARY OUTCOMES:
Collection from 3500 donors | Every six months

CONTACTS AND LOCATIONS:
Overall Officials: Janelle Cortner, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University Hospital, University of Lund, Malmo, Sweden

REFERENCES:
- [Background] Vermylen J. How do some haemophiliacs develop inhibitors? Haemophilia. 1998 Jul;4(4):538-42. doi: 10.1046/j.1365-2516.1998.440538.x. PMID 9873790
- [Background] Frommel D, Allain JP. Genetic predisposition to develop factor VIII antibody in classic hemophilia. Clin Immunol Immunopathol. 1977 Jul;8(1):34-8. doi: 10.1016/0090-1229(77)90089-7. No abstract available. PMID 880746
- [Background] Astermark J, Berntorp E, White GC, Kroner BL; MIBS Study Group. The Malmo International Brother Study (MIBS): further support for genetic predisposition to inhibitor development in hemophilia patients. Haemophilia. 2001 May;7(3):267-72. doi: 10.1046/j.1365-2516.2001.00510.x. PMID 11380630